CLINICAL TRIAL: NCT00746291
Title: Assessment of Autonomic Nervous System With Analysis of Heart Rate Variability in Children With Brain Damage.
Brief Title: Heart Rate Variability (HRV) Among Children With Brain Damage
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Alyn Pediatric & Adolescent Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: alyn3CTIL
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Brain Injury; Cerebral Palsy
MeSH Terms: conditions — Brain Injuries; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Traumatic brain injury
  Interventions: Other: 6 min walk test, Step climbing
- B (Experimental): Cerebral palsy
  Interventions: Other: 6 min walk test, Step climbing
- C (Experimental): Controls
  Interventions: Other: 6 min walk test, Step climbing

INTERVENTIONS:
Other: 6 min walk test, Step climbing — walking for 6 minute and climbing steps

SUMMARY:
to investigate the function of the autonomic nervous system in children with with post traumatic brain injury and children with cerebral palsy through an analysis of heart rate variability (HRV) occurring with walking performance.

DETAILED DESCRIPTION:
40 children with brain damage (20 with post TBI and 20 with CP)and 40 typically developed children will be participate in this study. ECG signals during rest and walking (for 6 minute and during step climbing) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* able to walk independently

Exclusion Criteria:

* can not follow simple commands

Ages: 6 Years to 12 Years | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
HRV parameters | during the assessment

CONTACTS AND LOCATIONS:
Overall Officials: Hemda Rotem, Principal Investigator — Alyn Hopspital Jerusalem
Locations (1):
- Alyn Pediatric and Adolescent Rehabilitation Center, Jerusalem, Israel